CLINICAL TRIAL: NCT07191041
Title: Emotional Distress in Recurrent Urinary Tract Infection
Brief Title: Emotional Urinary Tract Infection
Acronym: UTI
Status: Not yet recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bilal Chughtai, Chief of Urology, Northwell Health
Other Study IDs: IRB #: 24-0256
Record Dates: First submitted 2024-12-27; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Urinary Tract Infection(UTI); Recurrent Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Questionnaires to assess emotional distress: To assess the role laboratory results, have on psychological stress level and severity of bladder symptoms in female patients who presents with recurrent uncomplicated UTIs using patient-reported questionnaires (UTISA and PSS-10).

SUMMARY:
This project proposes a rigorous investigation into the psychological impact of positive urine culture results and recurrent urinary tract infections (UTIs) in women, with a particular focus on Interstitial Cystitis and Bladder Pain Syndrome patients. Interstitial cystitis (IC) or bladder pain syndrome (BPS) is a poorly understood chronic disorder that has an immense impact on quality of life. Stress has been demonstrated to exacerbate bladder symptoms in IC/BPS patients. Because it is often difficult to differentiate IC/BPS symptoms from UTIs, laboratory tests such as urine cultures are often obtained to rule out infectious etiology. Positive lab results can disrupt emotion regulation and impact a variety of health-related coping and outcomes. Chen et al demonstrated in a cohort of 57 IC/BPS patients that the pain index was associated with anxiety mood status and a tendency to develop a sense of hopelessness and helplessness. The impact of positive laboratory results has not been investigated in recurrent UTI patients. Identifying triggers for worsening urinary symptoms is important in the overall management of bladder symptoms therefore it is important to evaluate the impact positive lab results on psychosocial stress level in this population in order provide better patient counseling. By employing validated questionnaires and comprehensive assessments, the study aims to provide evidence-based recommendations for patient counseling and management strategies tailored to address emotional distress and symptom severity. The findings will contribute to improving the overall well-being and quality of life for women affected by recurrent UTIs and associated conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years of age
* Diagnosis of recurrent uncomplicated urinary tract infection (≥2 infections in 6 months or ≥3 infections in one year)
* Ability to complete questionnaires

Exclusion Criteria:

* Patients who had a urologic procedure in the last 3 months
* History of bladder malignancy
* History of exposure to pelvic radiation therapy
* Unwilling or unable to comply with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Females over the age of 18 years with recurrent uncomplicated UTIs.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2026-08-28 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Through study completion, an average of 1 year
  To assess the role laboratory results have on psychological stress level and severity of bladder symptoms in female patients who presents with recurrent uncomplicated UTIs by change in Urinary traction infection symptom assessment (UTISA) scores. The assessment is a 14-item instrument asking about the severity and bothersomeness of seven key uUTI symptoms. Lower score demonstrating less severity and bothersome UTI symptoms.

SECONDARY OUTCOMES:
Secondary Objective | Through study completion, an average of 1 year
  To determine if emotional distress scores is higher at baseline in IC/BPS compared to non-IC/BPS patients and if recurrent UTIs is exacerbates emotional distress more than non-IC/BPS patients by change in the Perceived Stress scale (PSS-10) scores. Total score can range from 0 to 40. Lower score indicate lower perceived stress levels.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Northwell Health
Locations (1):
- NHPP Urology, Syosset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared as supplementary material accompanying the publication of the study results.

REFERENCES:
- [Background] Stanford E, McMurphy C. There is a low incidence of recurrent bacteriuria in painful bladder syndrome/interstitial cystitis patients followed longitudinally. Int Urogynecol J Pelvic Floor Dysfunct. 2007 May;18(5):551-4. doi: 10.1007/s00192-006-0184-9. Epub 2006 Oct 12. PMID 17036170
- [Background] Cihan A, Cihan E, Çakmak B. Perceived Stress and Accompanying Low Urine pH Are in Relation to Bladder Pain Syndrome. Journal of Urological Surgery. 2021;8:98-105.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Clayson D, Wild D, Doll H, Keating K, Gondek K. Validation of a patient-administered questionnaire to measure the severity and bothersomeness of lower urinary tract symptoms in uncomplicated urinary tract infection (UTI): the UTI Symptom Assessment questionnaire. BJU Int. 2005 Aug;96(3):350-9. doi: 10.1111/j.1464-410X.2005.05630.x. PMID 16042729
- [Background] Chen W-C, Lee M-H, Wu H-C. Relationship among symptoms, mood, and personality traits in patients with interstitial cystitis/bladder pain syndrome. Urological Science. 2017;28(3):147-151.
- [Background] Koziol JA, Clark DC, Gittes RF, Tan EM. The natural history of interstitial cystitis: a survey of 374 patients. J Urol. 1993 Mar;149(3):465-9. doi: 10.1016/s0022-5347(17)36120-7. PMID 8437248